CLINICAL TRIAL: NCT03381560
Title: An Observational, Cross-sectional Study of Primary Data Collection to Describe Symptoms Over 24 Hours and Their Relationship With Adherence to Respiratory Treatment, Direct Costs and PRO in Stable COPD Patients in Brazil.
Brief Title: A Study to Evaluate the Symptoms Over 24 Hours in Patients With Chronic Obstructive Pulmonary Disease - LASSYC Study
Acronym: LASSYC
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00119
Record Dates: First submitted 2017-12-18; First posted 2017-12-22 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: LASSYC; COPD symptoms.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
No previous studies have evaluated the frequency and severity of Chronic Obstructive Pulmonary Disease (COPD) symptoms over a period of 24 hours (early morning, daytime and nigth-time symptoms) in stable COPD patients seen in clinical practice in Brazil. COPD is a common disease seen by primary care physicians and one of the most common diseases referred and diagnosed by pulmonologists. According to previous studies, symptoms of COPD can have a substantial impact on patients' quality of life and present a considerable degree of variation for the same degree of airflow limitation.

The objective of this study is to learn more about the burden of symptoms in the real-world population of COPD patients in Brazil. With the real life data coming from this study, it will be possible to describe 24-hour COPD symptoms in Brazil and their impact on patients' quality of life and other PROs, the relationship with patients´ behaviour regarding adherence to respiratory medication and burden of COPD symptoms in terms of the impact on health economics.

In the present study, the investigators will assess and characterize COPD symptoms over a period of 24 hours, by collecting information about the respiratory symptoms experienced at different times of the day and night in patients with stable COPD under real clinical practice conditions. In addition, the investigators will evaluate the correlation between each of these symptoms and the GOLD classification, adherence to respiratory treatment, level of dyspnea, disease severity, comorbidities and physical activity. Finally, the investigators will assess the relationship between 24h symptoms and direct cost related to treatment and HRU in the previous year to assess the burden of COPD symptoms.

The present study is based on a similar protocol applied in Latin-American patients, the LASSYC Study. Extracted data will be used for a Brazilian analysis of these outcomes and may be used in future analyses combined with the results of LASSYC Study for a global view of Latin America.

DETAILED DESCRIPTION:
Background

Chronic Obstructive Pulmonary Disease (COPD) is a preventable and treatable disease with some significant extrapulmonary effects that may contribute to the severity in individual patients. Its pulmonary component is characterized by airflow limitation that is not fully reversible. The airflow limitation is usually progressive and associated with an abnormal inflammatory response of the lung to noxious particles or gases (i). Although smoking is one of the major and most frequent causes of COPD, other factors may be associated with its development. The narrowing of the airways, which is one of the main features of COPD, results from a combination of small airway disease and parenchymal destruction, as well as structural changes from the chronic inflammatory process. For this reason bronchoconstriction is one of the key targets of pharmacological interventions in the management of COPD.

This disease affects globally around 15% of all adults older than 40 years, resulting in pulmonary and extrapulmonary comorbidities and significant mortality (1,ii). The worldwide prevalence in people aged over 40 years is 10.1% overall, 11.8% for men, and 8.5% for women, according to the BOLD Study (iii). It is the fourth leading cause of death in the world and its prevalence is projected to increase in the coming years due to continued exposure to COPD risk factors (1). Two Latin-American epidemiological studies, the PLATINO Project iv and PREPOCOL v, have provided information on the prevalence of COPD in this region. PLATINO is a study on prevalence of COPD in individuals ≥40 years, carried out in five Latin American cities: Mexico City (Mexico), São Paulo (Brazil), Montevideo (Uruguay), Santiago de Chile (Chile), and Caracas (Venezuela). Using as diagnostic criteria post-BD FEV1/FVC ratio <0.70, the overall prevalence of COPD in PLATINO is 14.3% (ranging from 7.8% in Mexico City to 19.7% in Montevideo) and in the city of São Paulo is 15.8 % (4,vi). Using the lower limit of normal criteria (LLN) of the post- BD FEV1/FVC ratio, the global COPD prevalence in PLATINO is 11.7%. This is even lower (9.5%) when using the post-BD FEV1/VEF6 < LLN ratio (vii). PREPOCOL (5) assessed the prevalence in five cities in Colombia and reported an overall prevalence of 8.9% (from 6.2% in Barranquilla to 13,5% in Medellin).

Symptoms of COPD - including progressive dyspnea, chronic cough, excessive sputum production and decreased exercise tolerance - may considerably affect the patients' daily activities and quality of life (1,viii,ix). COPD symptoms have been reported to be worse at night and in the early morning (x,xi), which may be reflected in disturbed sleep and limitations on morning activities.

Moreover, the health-related quality of life (HRQoL) is being recognized as an important outcome when evaluating patients with COPD and several studies have demonstrated that those patients in more severe disease stages presented worse HRQoL and it varied greatly within each stage of disease severity (xii).

From the patient´s point of view, dyspnea is one of the major symptoms that affect their quality of life (xiii). However, dyspnea varies considerably for the same degree of airflow limitation.

It is reported that poor patient's adherence to inhaled medication is shared by COPD and asthma patients (xiv). Non-adherence to inhaled therapy is associated with inadequate symptom control, higher healthcare utilization and costs, as well as decreases in health-related quality of life (12- 14). In practice guidelines of the Global Initiative for Asthma Management [GINA) (xv) and Global Initiative for Chronic Obstructive Lung Disease (GOLD) (1)] is now specifically recommended evaluation and follow-up of the patient's adherence to inhaler devices.

Previous studies (xvi, xvii, xviii, xix) have shown that physical activity in COPD is associated with a better quality of life and less morbidity and mortality. In addition, comorbid conditions such as cardiovascular disease, anxiety and depressive disorders, lung cancer and osteoporosis are frequently observed in COPD patients and may affect COPD outcomes (xx). Sleep disorder is also common in COPD patients. In epidemiologic studies, more than 50% of patients with COPD complained of difficulty to maintain and initiate sleep, and 25% complained of excessive daytime sleepiness (xxi). The COTE Index establishes the relationship between these main comorbidities and the risk of death over a median of 51 months. This is a simple, disease-specific comorbidity index that helps assess the risk of mortality in patients with COPD (xxii).

It has been recently published the ASSESS Study (xxiii) regarding a cohort of 727 European patients. This observational study assessed the prevalence, severity and relationship between nighttime, early morning and daytime COPD symptoms and explored the relationship between 24-hour symptoms and other results reported by DPOC patients. It was shown that more than half of patients experienced COPD symptoms throughout the whole 24-hour period, and there was a significant relationship between them and the worse patient-reported outcome, suggesting that improving 24- hour symptoms should be an important consideration in the management of COPD.

COPD is associated with a substantial economic burden due to direct healthcare costs e.g. unplanned medical visits and hospitalization due to exacerbations (1,xxiv). More frequent exacerbations are associated with: more frequent/longer hospital stays; increased mortality risk; reduced quality of life (xxv); as well as indirect/societal costs due to loss of productivity and premature death in patients with COPD further increasing the economic burden of this disease (1,24-xxvi).

Rationale

No previous studies have evaluated the frequency and severity of COPD symptoms over a period of 24 hours (nighttime, early morning and daytime symptoms) in stable COPD patients seen in clinical practice in Brazil. COPD is a common disorder seen by primary care physicians and one of the most common diseases referred and diagnosed by pulmonologists. According to studies, COPD symptoms can have a substantial impact on patients' quality of daily life and present a considerable degree of variation for the same degree of airflow limitation.

This study aims to learn more about the burden of symptoms in the real-world population of COPD patients in Brazil. With the real life data from this study, it will be possible to describe 24-hour COPD symptoms and their impact on patients' quality of life and other PRO, the relationship with patients' behaviour regarding adherence to respiratory medication and the burden of COPD symptoms in terms of the impact on health economics in Brazil.

In the present study, the investigators will assess and characterize COPD symptoms over a period of 24 hours, by collecting information about the respiratory symptoms experienced at different times of the day and night-time in patients with stable COPD under real clinical practice conditions. In addition, the investigators will evaluate the correlation between each of these symptoms and the 2013 GOLD classification, adherence to respiratory treatment, level of dyspnea, disease severity, comorbidities and physical activity. Finally, the investigators will assess the relationship between 24h symptoms and direct cost related to treatment and HRU in the previous year to assess the burden of COPD symptoms.

ELIGIBILITY:
INCLUSION CRITERIA

Patients will only be included in the study if they meet all of the following criteria:

1. Male or female patients aged 40 years or older.
2. Patient diagnosed with COPD for 1 year or more.
3. Patient presenting at least one spirometry with COPD criteria, FEV1/FVC fixed ratio <0.70 post BD, in the last 12 months.
4. Patient is a current smoker or an ex-smoker with a smoking history of ≥ 10 pack- years.
5. Stable patients, as stated in medical records or patient reports during visit, defined as: without treatment due to exacerbation at study visit or within the previous 2 months, and without changes in maintenance COPD treatment regimen over the preceding 2 months (avoid first-time patient from participating in the study).
6. Patients must be able and willing to read and understand written instructions, and understand and complete the questionnaires required by the protocol.
7. After receiving full explanation, patients must have signed an informed consent document indicating that they understand the purpose of and the procedures required for the study and are willing to participate in the study.

EXCLUSION CRITERIA

Patients who meet any of the following criteria will not be eligible to participate in the study:

1. Patient with a diagnosis of sleep apnea syndrome or other chronic respiratory disease different from chronic obstructive diseases.
2. An acute or chronic condition that, in the investigator's opinion, would limit patient's ability to complete the questionnaires or participate in this study.

Ages: 40 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of 40 years and older, smokers or ex smokers of >= 10 pack/years with previous COPD diagnosis, attending outpatient specialists consults in Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Frequency of COPD-related nighttime symptoms | 24 hours
Mean severity of COPD-related nighttime symptoms | 24 hours
Frequency of COPD-related daytime symptoms | 24 hours
Mean severity of COPD-related daytime symptoms | 24 hours
Frequency of COPD-related early morning symptoms | 24 hours
Mean severity of COPD-related early morning symptoms | 24 hours
Interrelationship between early morning, day and nighttime symptoms | 24 hours

SECONDARY OUTCOMES:
Relationship between early morning, day and nighttime symptoms and adherence to respiratory medication. | 6 months
Relationship between early morning, day and nighttime symptoms and disease classification (GOLD 2013) | 6 months
Relationship between early morning, day and nighttime symptoms and disease severity and prognostic assessment (BODEx) | 6 months
Relationship between early morning, day and nighttime symptoms and level of dyspnea (mMRC) | 6 months
Relationship between early morning, day and nighttime symptoms and HRQoL (CAT) | 6 months
Relationship between early morning, day and nighttime symptoms and presence of comorbidities (COTE) | 6 months
Relationship between early morning, day and nighttime symptoms and history of exacerbations within the past 12 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Cukier, Principal Investigator — Instituto do Coração do Hospital das Clínicas da FMUSP
Locations (7):
- Brazil (7):
  - Research Site, Blumenau
  - Research Site, Botucatu
  - Research Site, Campinas
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São Bernardo do Campo
  - Research Site, São Paulo

REFERENCES:
- [Derived] Cukier A, Godoy I, Costa CHD, Rubin AS, Gregorio MG, Albuquerque Neto AA, Lima MA, Pereira MC, Tanni SE, Athanazio RA, Bessa EJC, Wehrmeister FC, Lourenco CB, Menezes AMB. Symptom variability over the course of the day in patients with stable COPD in Brazil: a real-world observational study. J Bras Pneumol. 2019 Dec 20;46(3):e20190223. doi: 10.36416/1806-3756/e20190223. eCollection 2020. PMID 31859705
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2287R00119&attachmentIdentifier=b2616b0f-2fec-4c38-90b9-a3d5851ecab7&fileName=LASSYC-BR_CSR_Synopsis_D2287R00119_26June2019.pdf&versionIdentifier=